CLINICAL TRIAL: NCT04358835
Title: Keto-diet for Intubated Critical Care COVID-19 (KICC-COVID19)
Brief Title: Keto-diet for Intubated Critical Care COVID-19
Acronym: KICC-COVID19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not begin enrollment, multiple competing studies at same institution
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00247383
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: COVID-19
Keywords: ketogenic diet; Intensive care; COVID-19; Mechanical ventilation; Intubated patients; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Diet, Ketogenic; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a single-center, open-label, clinical trial designed to determine whether a ketogenic diet improves gas exchange and reduces ventilator requirements in patients with coronavirus disease intubated for respiratory failure. The study team will prospectively enroll 15 intubated patients with COVID-19 infection and administer a 4:1 ratio enteral ketogenic formula within 48 hours of intubation. This study will compare outcomes to a retrospective cohort of intubated patients with COVID-19 who did not receive ketogenic diet. As other clinical trials begin, co-administration of other therapies as well as standard care treatments will be recorded. In addition, the study will compare clinical outcomes with patients receiving exclusively standard clinical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intubated patients with COVID-19 on a ketogenic diet only (Experimental): 4:1 ketogenic diet formula
  Interventions: Dietary Supplement: Ketogenic diet; Other: standard of care

INTERVENTIONS:
Dietary Supplement: Ketogenic diet — 4:1 ratio enteral ketogenic formula within 48 hours of intubation
Other: standard of care — standard of care/supportive therapy

SUMMARY:
Coronavirus disease (COVID-2019) is a devastating viral illness that originated in Wuhan China in late 2019 and there are nearly 2 million confirmed cases. The mortality rate is approximately 5% of reported cases and over half of patients that require mechanical ventilation for respiratory failure. As the disease continues to spread, strategies for reducing duration of ventilator support in patients with COVID-19 could significantly reduce morbidity and mortality of these individuals and future patients requiring this severely limited life-saving resource. Methods to improve gas exchange and to reduce the inflammatory response in COVID-19 are desperately needed to save lives.

The ketogenic diet is a high fat, low carbohydrate, adequate-protein diet that promotes metabolic ketosis (ketone body production) through hepatic metabolism of fatty acids. High fat, low carbohydrate diets have been shown to reduce duration of ventilator support and partial pressure carbon dioxide in patients with acute respiratory failure. In addition, metabolic ketosis reduces systemic inflammation. This mechanism could be leveraged to halt the cytokine storm characteristic of COVID-19 infection.

The hypothesis of this study is that the administration of a ketogenic diet will improve gas exchange, reduce inflammation, and duration of mechanical ventilation. The plan is to enroll 15 intubated patients with COVID 19 infection and administer a 4:1 ketogenic formula during their intubation.

DETAILED DESCRIPTION:
Coronavirus disease (COVID-2019) is a devastating viral illness that originated in Wuhan China in late 2019. The number of confirmed cases worldwide has nearly reached 2 million and more than 125,000 people have died. Early studies from Wuhan reported a mortality rate of 2-3% with lower rates in surrounding provinces as the disease spread (closer to 0.7% of confirmed cases). One hypothesized cause for the higher mortality rate in Wuhan compared to surrounding regions was the rapid "surge" of COVID-19 infections before the disease was identified and social distancing implemented. Critically ill patients developed acute respiratory distress syndrome with inflammatory pulmonary edema and life-threatening hypoxemia requiring mechanical ventilation. This resulted in a significant strain on health-care resources such as availability of mechanical ventilators to treat patients with acute respiratory failure. As the disease spreads worldwide, strategies for reducing duration of ventilator support in patients with COVID-19 could significantly reduce morbidity and mortality of these individuals and future patients requiring this severely limited life-saving resource.

Alterations in macronutrient composition may be leveraged to improve ventilation and inflammation in COVID-19 patients. The ketogenic diet is a high fat, low carbohydrate, adequate protein diet that promotes ketone body production through hepatic metabolism of fatty acids. High fat, low carbohydrate diets have been shown to reduce duration of ventilator support and partial pressure carbon dioxide in patients with acute respiratory failure. Switching from glucose to fat oxidation lowers the respiratory quotient, thereby reducing the amount of carbon dioxide produced. This reduces ventilator demands and may improve oxygenation by lowering alveolar carbon dioxide levels, ultimately reducing time on mechanical ventilation. A study published in 1989 compared 10 participants intubated for acute respiratory failure and randomized to a high-fat, low carbohydrate diet and 10 participants receiving a standard isocaloric, isonitrogenous diet and showed a decrease in the partial pressure of carbon dioxide of 16% in the ketogenic diet group compared to a 4% increase in the standard diet group (p=0.003). The patients in the high-fat diet group had a mean of 62 fewer hours on a ventilator (p = 0.006) compared to the control group.

The high-fat diet used in the study had a ratio of 1.2:1 fat to protein and carbohydrate combined in grams. The ketogenic diet, which has been used safely and effectively in patients with chronic epilepsy for nearly one century and more recently in critically ill, intubated patients for the management of refractory and super-refractory status epilepticus has a 4:1 ratio (90% fat kilocalories). While a 1:1 ratio diet can produce a state of mild metabolic ketosis (typically ~ 1 mmol/L of the ketone body betahydroxybutyrate, measured in serum), a higher 4:1 ratio ketogenic diet can produce higher ketone body betahydroxybutyrate levels and more rapidly (up to 2 mmol/L within 24 hours of initiation). One study of obese patients treated with ketogenic diet reported that increases in ketone body production correlated with a lower partial pressure of carbon dioxide levels. A more recent study showed that patients with refractory epilepsy had a reduction in the respiratory quotient and increased fatty acid oxidation without a change in the respiratory energy expenditure with chronic use of the ketogenic diet. These findings were replicated in healthy subjects on ketogenic diet compared to a control group and patients on a ketogenic diet also had a significant reduction in carbon dioxide output and partial pressure of carbon dioxide. The authors concluded that a ketogenic diet may decrease carbon dioxide body stores and that use of a ketogenic diet may be beneficial for patients with respiratory failure. Even in patients without hypercapnia (primarily hypoxic respiratory failure), lowering carbon dioxide production permits lowering tidal volumes - a cornerstone of acute respiratory distress syndrome management.

In addition to reducing the partial pressure of carbon dioxide, metabolic ketosis reduces systemic inflammation. This mechanism could be leveraged to halt the cytokine storm characteristic of COVID-19 infection. Several studies provide evidence that pro-inflammatory cytokine production is significantly reduced in animals fed a ketogenic diet in a variety of disease models. In a rodent model of Parkinson's disease, mice were found to have significantly decreased levels of pro-inflammatory, macrophage secreted cytokines interleukin-1β, interleukin-6, and Tumor necrosis factor-alpha after 1 week of treatment with a ketogenic diet. Likewise, rats pretreated with a ketogenic diet prior to injection with lipopolysaccharide to induce fever did not experience an increase in body temperature or interleukin-1β, while significant increases were seen in control animals not pretreated with a ketogenic diet. In a mouse model of NLRP3-mediated diseases as well as human monocytes, the ketone body beta-hydroxybutyrate inhibited the NLRP3 inflammasome-mediated production of interleukin-1β and interleukin-18. These findings have been replicated in several recent animal studies and preliminary studies in humans. The hypothesis of this study is that through induction of metabolic ketosis combined with carbohydrate restriction, a ketogenic diet is protective against the cytokine storm in COVID-19. With its carbon dioxide-lowering and anti-inflammatory properties, a ketogenic diet may become an important component of the acute respiratory distress syndrome arsenal with immediate relevance to the current COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older.
* COVID-19 positive and respiratory failure requiring intubation
* Legally authorized representative

Exclusion Criteria:

* Unstable metabolic condition
* Liver failure
* Acute Pancreatitis
* Inability to tolerate enteral feeds, ileus, gastrointestinal bleeding
* Known Pregnancy
* Received propofol infusion within 24 hours
* Known fatty acid oxidation disorder or pyruvate carboxylase deficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the partial pressure of carbon dioxide (PaCO2) | Daily until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  PaCO2 is the partial pressure of carbon dioxide Units: millimeters of mercury

SECONDARY OUTCOMES:
Change in minute ventilation | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Minute ventilation is the product of respiratory rate and tidal volume. Units: Liter per minute
Change in respiratory system compliance | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Respiratory system compliance measures the extent to which the lungs will expand.
  In a ventilated patient, compliance can be measured by dividing the delivered tidal volume by the [plateau pressure minus the total peep]. Units: liter/centimeter of water
Change in driving pressure | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Driving pressure is a measure of the strain applied to the respiratory system and the risk of ventilator-induced lung injuries Driving pressure = Plateau pressure - Total Positive end-expiratory pressure (PEEP) Units: centimeter of water
Change in ventilator synchrony | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Ventilator synchrony is the match between the patient's neural inspiratory time and the ventilator insufflation time
Change in mean arterial pressure | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Mean arterial pressure is the average pressure in a patient's arteries during one cardiac cycle. Mean arterial pressure = diastolic blood pressure +[1/3(systolic blood pressure - diastolic blood pressure)] Units: millimeter of mercury
Change in the fraction of inspired oxygen percentage of oxygen (FiO2) | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  FiO2: Fraction of Inspired Oxygen Percentage of oxygen in the air mixture that is delivered to the patient.
  Units: %
Change in the partial pressure of carbon dioxide (PaO2) to the fraction of inspired oxygen percentage of oxygen (FiO2) ratio | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  PaO2/FiO2 ratio is the ratio of arterial oxygen partial pressure (PaO2) to fractional inspired oxygen.
  Units: millimeter of mercury
Change in hydrogen ion activity (pH) | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  pH measures hydrogen ion activity. It is a conventional part of every arterial blood gas determination pH: no units.
Change in Bicarbonate (HCO3) | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Bicarbonate is a conventional part of every arterial blood gas determination Units: milliequivalents/Liter
Change in red blood cell count | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Red blood cell count measure anemia or hypoglycemia. Units: cells per liter
Change in white blood cell count | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  White blood cell count evaluates leukopenia or leukocytosis. Units: cells/liter
Change in white cell differential | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  White cell differential shows the amount of neutrophils, lymphocytes, basophils, eosinophils and may give some clue of the type of infection. Units: %
Change in hemoglobin levels | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Hemoglobin is an indirect way to measure red blood cells. Units: gram/deciliter
Change in hematocrit | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Hematocrit measures the volume percentage of red blood cells in blood. Units: %
Change in mean cell volume | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Mean cell volume is a measure of the average volume of a red blood corpuscle. Units: femtoliters
Change in mean cell hemoglobin | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Mean cell hemoglobin is the average mass of hemoglobin per red blood cell in a sample of blood. Units: picograms
Change in mean cell hemoglobin concentration | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Mean cell hemoglobin concentration is the average concentration of hemoglobin in a given volume of blood. Units: %
Change in platelet count | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Platelet count measures the number of platelets in the blood and determines thrombocytopenia or thrombocytosis. Units: platelets/liter
Change in red cell distribution width | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Red cell distribution width is a measure of the range of variation of red blood cell volume. Units: no units
Change in blood albumin level | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Liver function test Units: gram/deciliter
Change in serum alkaline phosphatase level | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Liver function test Units: international units/liter
Change in serum aspartate transaminase level | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Liver function test Units: international units/liter
Change in serum alanine aminotransferase level | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Liver function test Units: international units/liters
Change in blood urea nitrogen levels | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Kidney function test Units: milligram/deciliter
Change in serum calcium level | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Kidney function test Units: milligram/deciliter
Change in serum chloride level | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Kidney function test Units: millimole/liter
Change in serum potassium level | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Kidney function test Units: millimole/liter
Change in serum creatinine level | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Kidney function test Units: gram/deciliter
Date patient is re-intubated or need mechanical ventilation for a second time | Up to 10 days
  If the patient needs mechanical ventilation for a second time, this information will be collected.
Length of intensive care unit stay | Up to 10 days
  Time from intensive care unit admission until death or transfer to hospital bed.
The total hospital stay | Up to 10 days
  Time from hospital admission to discharge from the hospital. This information will be collected.
Disposition at discharge | Up to 10 days
  Once the patient feels better and can leave the hospital, he/she will be discharged. The place of discharge (e.g. home, rehab facility, nursing home, etc), time and date will be collected.
Change in heart rate | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Heart rate: is the number of times a person's heart beats per minute
Change in the dosage of vasopressor medication | every 6 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Units: milligram

OTHER OUTCOMES:
Change in total blood cholesterol level | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Units: milligram/deciliter
Change in blood low-density lipoprotein level | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Units: milligram/deciliter
Change in blood high-density lipoprotein level | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Units: milligram/deciliter
Change in blood triglycerides level | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Units: milligram/deciliter
Change in blood glucose level | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Glucose: sugar in blood. Units: millimole/liter
Change in blood glucagon level | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Glucagon: hormone release by pancreas that increase concentration of glucose in blood. Units: nanogram/liter
Change in blood free fatty acids level | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Free fatty acids are fatty acids that are produced from triglycerides and are measure in blood.
Change in blood insulin levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Hormone that regulates glucose. Units: insulin units/liter
Change in blood leptin levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Leptin helps regulate and alter long-term food intake and energy expenditure. Units: nanogram/deciliter
Change in blood insulin like growth factor 1 levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Units: nanomole/liter
Change in blood C-reactive protein levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  C-reactive protein is a protein made by the liver that measures inflammation (e.g. pancreatitis). Units: microgram/milliliter
Change in blood interleukin-1β levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Cytokines are signaling molecules that measure inflammation.
Change in blood interleukin-6 levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Cytokines are signaling molecules that measure inflammation.
Change in blood interleukin-18 levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Cytokines are signaling molecules that measure inflammation.
Change in blood tumor necrosis factor alpha levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Cytokines are signaling molecules that measure inflammation.
Change in blood C-C motif chemokine ligand 2 (CCL2) levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Chemokine that mediates inflammation.
Change in blood C-C motif chemokine ligand 3 (CCL3) levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Chemokine that mediates inflammation.
Change in blood C-C motif chemokine ligand 4 (CCL4) levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Chemokine that mediates inflammation.
Change in blood B cell-attracting chemokine 1 (CXCL13) levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Chemokine that mediates inflammation.
Change in blood ferritin levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Ferritin stores iron inside of cells. Units: nanogram/milliliter
Change in blood betahydroxybutyrate levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Units: millimole/liter
Change in blood urine acetoacetate levels | At baseline and every 24 hours until the patient is wean off the ventilator or die, whichever came first, assessed up to 10 days
  Units: millimole/liter

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie Cervenka, MD, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Background] Ji Y, Ma Z, Peppelenbosch MP, Pan Q. Potential association between COVID-19 mortality and health-care resource availability. Lancet Glob Health. 2020 Apr;8(4):e480. doi: 10.1016/S2214-109X(20)30068-1. Epub 2020 Feb 25. No abstract available. PMID 32109372
- [Background] al-Saady NM, Blackmore CM, Bennett ED. High fat, low carbohydrate, enteral feeding lowers PaCO2 and reduces the period of ventilation in artificially ventilated patients. Intensive Care Med. 1989;15(5):290-5. doi: 10.1007/BF00263863. PMID 2504796
- [Background] van den Berg B, Bogaard JM, Hop WC. High fat, low carbohydrate, enteral feeding in patients weaning from the ventilator. Intensive Care Med. 1994 Aug;20(7):470-5. doi: 10.1007/BF01711897. PMID 7995861
- [Background] Cervenka MC, Hartman AL, Venkatesan A, Geocadin RG, Kossoff EH. The ketogenic diet for medically and surgically refractory status epilepticus in the neurocritical care unit. Neurocrit Care. 2011 Dec;15(3):519-24. doi: 10.1007/s12028-011-9546-3. PMID 21523523
- [Background] Cervenka MC, Hocker S, Koenig M, Bar B, Henry-Barron B, Kossoff EH, Hartman AL, Probasco JC, Benavides DR, Venkatesan A, Hagen EC, Dittrich D, Stern T, Radzik B, Depew M, Caserta FM, Nyquist P, Kaplan PW, Geocadin RG. Phase I/II multicenter ketogenic diet study for adult superrefractory status epilepticus. Neurology. 2017 Mar 7;88(10):938-943. doi: 10.1212/WNL.0000000000003690. Epub 2017 Feb 8. PMID 28179470
- [Background] McDonald TJW, Cervenka MC. Ketogenic Diets for Adults With Highly Refractory Epilepsy. Epilepsy Curr. 2017 Nov-Dec;17(6):346-350. doi: 10.5698/1535-7597.17.6.346. PMID 29217974
- [Background] Williams TJ, Cervenka MC. The role for ketogenic diets in epilepsy and status epilepticus in adults. Clin Neurophysiol Pract. 2017 Jul 1;2:154-160. doi: 10.1016/j.cnp.2017.06.001. eCollection 2017. PMID 30214989
- [Background] Thakur KT, Probasco JC, Hocker SE, Roehl K, Henry B, Kossoff EH, Kaplan PW, Geocadin RG, Hartman AL, Venkatesan A, Cervenka MC. Ketogenic diet for adults in super-refractory status epilepticus. Neurology. 2014 Feb 25;82(8):665-70. doi: 10.1212/WNL.0000000000000151. Epub 2014 Jan 22. PMID 24453083
- [Background] McDonald TJW, Henry-Barron BJ, Felton EA, Gutierrez EG, Barnett J, Fisher R, Lwin M, Jan A, Vizthum D, Kossoff EH, Cervenka MC. Improving compliance in adults with epilepsy on a modified Atkins diet: A randomized trial. Seizure. 2018 Aug;60:132-138. doi: 10.1016/j.seizure.2018.06.019. Epub 2018 Jun 22. PMID 29960852
- [Background] Park EG, Lee J, Lee J. The ketogenic diet for super-refractory status epilepticus patients in intensive care units. Brain Dev. 2019 May;41(5):420-427. doi: 10.1016/j.braindev.2018.12.007. Epub 2019 Jan 9. PMID 30638692
- [Background] Peng P, Peng J, Yin F, Deng X, Chen C, He F, Wang X, Guang S, Mao L. Ketogenic Diet as a Treatment for Super-Refractory Status Epilepticus in Febrile Infection-Related Epilepsy Syndrome. Front Neurol. 2019 Apr 26;10:423. doi: 10.3389/fneur.2019.00423. eCollection 2019. PMID 31105638
- [Background] Fried PI, McClean PA, Phillipson EA, Zamel N, Murray FT, Marliss EB. Effect of ketosis on respiratory sensitivity to carbon dioxide in obesity. N Engl J Med. 1976 May 13;294(20):1081-6. doi: 10.1056/NEJM197605132942003. PMID 1256524
- [Background] Tagliabue A, Bertoli S, Trentani C, Borrelli P, Veggiotti P. Effects of the ketogenic diet on nutritional status, resting energy expenditure, and substrate oxidation in patients with medically refractory epilepsy: a 6-month prospective observational study. Clin Nutr. 2012 Apr;31(2):246-9. doi: 10.1016/j.clnu.2011.09.012. Epub 2011 Oct 20. PMID 22019282
- [Background] Rubini A, Bosco G, Lodi A, Cenci L, Parmagnani A, Grimaldi K, Zhongjin Y, Paoli A. Effects of Twenty Days of the Ketogenic Diet on Metabolic and Respiratory Parameters in Healthy Subjects. Lung. 2015 Dec;193(6):939-45. doi: 10.1007/s00408-015-9806-7. Epub 2015 Sep 26. PMID 26410589
- [Background] Ruskin DN, Ross JL, Kawamura M Jr, Ruiz TL, Geiger JD, Masino SA. A ketogenic diet delays weight loss and does not impair working memory or motor function in the R6/2 1J mouse model of Huntington's disease. Physiol Behav. 2011 Jul 6;103(5):501-7. doi: 10.1016/j.physbeh.2011.04.001. Epub 2011 Apr 9. PMID 21501628
- [Background] Yang X, Cheng B. Neuroprotective and anti-inflammatory activities of ketogenic diet on MPTP-induced neurotoxicity. J Mol Neurosci. 2010 Oct;42(2):145-53. doi: 10.1007/s12031-010-9336-y. Epub 2010 Mar 24. PMID 20333481
- [Background] Fraser DA, Thoen J, Bondhus S, Haugen M, Reseland JE, Djoseland O, Forre O, Kjeldsen-Kragh J. Reduction in serum leptin and IGF-1 but preserved T-lymphocyte numbers and activation after a ketogenic diet in rheumatoid arthritis patients. Clin Exp Rheumatol. 2000 Mar-Apr;18(2):209-14. PMID 10812493
- [Background] Fraser DA, Thoen J, Djoseland O, Forre O, Kjeldsen-Kragh J. Serum levels of interleukin-6 and dehydroepiandrosterone sulphate in response to either fasting or a ketogenic diet in rheumatoid arthritis patients. Clin Exp Rheumatol. 2000 May-Jun;18(3):357-62. PMID 10895373
- [Background] Schreck KC, Lwin M, Strowd RE, Henry-Barron BJ, Blakeley JO, Cervenka MC. Effect of ketogenic diets on leukocyte counts in patients with epilepsy. Nutr Neurosci. 2019 Jul;22(7):522-527. doi: 10.1080/1028415X.2017.1416740. Epub 2017 Dec 18. PMID 29254457
- [Background] Chen C, Zhang XR, Ju ZY, He WF. [Advances in the research of mechanism and related immunotherapy on the cytokine storm induced by coronavirus disease 2019]. Zhonghua Shao Shang Za Zhi. 2020 Jun 20;36(6):471-475. doi: 10.3760/cma.j.cn501120-20200224-00088. Chinese. PMID 32114747
- [Background] Buyken AE, Goletzke J, Joslowski G, Felbick A, Cheng G, Herder C, Brand-Miller JC. Association between carbohydrate quality and inflammatory markers: systematic review of observational and interventional studies. Am J Clin Nutr. 2014 Apr;99(4):813-33. doi: 10.3945/ajcn.113.074252. Epub 2014 Feb 19. PMID 24552752
- [Background] Dupuis N, Curatolo N, Benoist JF, Auvin S. Ketogenic diet exhibits anti-inflammatory properties. Epilepsia. 2015 Jul;56(7):e95-8. doi: 10.1111/epi.13038. Epub 2015 May 23. PMID 26011473
- [Background] Youm YH, Nguyen KY, Grant RW, Goldberg EL, Bodogai M, Kim D, D'Agostino D, Planavsky N, Lupfer C, Kanneganti TD, Kang S, Horvath TL, Fahmy TM, Crawford PA, Biragyn A, Alnemri E, Dixit VD. The ketone metabolite beta-hydroxybutyrate blocks NLRP3 inflammasome-mediated inflammatory disease. Nat Med. 2015 Mar;21(3):263-9. doi: 10.1038/nm.3804. Epub 2015 Feb 16. PMID 25686106
- [Background] Bae HR, Kim DH, Park MH, Lee B, Kim MJ, Lee EK, Chung KW, Kim SM, Im DS, Chung HY. beta-Hydroxybutyrate suppresses inflammasome formation by ameliorating endoplasmic reticulum stress via AMPK activation. Oncotarget. 2016 Oct 11;7(41):66444-66454. doi: 10.18632/oncotarget.12119. PMID 27661104
- [Background] Deora V, Albornoz EA, Zhu K, Woodruff TM, Gordon R. The Ketone Body beta-Hydroxybutyrate Does Not Inhibit Synuclein Mediated Inflammasome Activation in Microglia. J Neuroimmune Pharmacol. 2017 Dec;12(4):568-574. doi: 10.1007/s11481-017-9754-5. Epub 2017 Aug 23. PMID 28836226
- [Background] Goldberg EL, Asher JL, Molony RD, Shaw AC, Zeiss CJ, Wang C, Morozova-Roche LA, Herzog RI, Iwasaki A, Dixit VD. beta-Hydroxybutyrate Deactivates Neutrophil NLRP3 Inflammasome to Relieve Gout Flares. Cell Rep. 2017 Feb 28;18(9):2077-2087. doi: 10.1016/j.celrep.2017.02.004. PMID 28249154
- [Background] Yamanashi T, Iwata M, Kamiya N, Tsunetomi K, Kajitani N, Wada N, Iitsuka T, Yamauchi T, Miura A, Pu S, Shirayama Y, Watanabe K, Duman RS, Kaneko K. Beta-hydroxybutyrate, an endogenic NLRP3 inflammasome inhibitor, attenuates stress-induced behavioral and inflammatory responses. Sci Rep. 2017 Aug 9;7(1):7677. doi: 10.1038/s41598-017-08055-1. PMID 28794421
- [Background] Baumeister FA, Oberhoffer R, Liebhaber GM, Kunkel J, Eberhardt J, Holthausen H, Peters J. Fatal propofol infusion syndrome in association with ketogenic diet. Neuropediatrics. 2004 Aug;35(4):250-2. doi: 10.1055/s-2004-820992. PMID 15328567
- [Background] Brozova K, Broz J. The risk of hypoglycemia and the ketogenic diet for super-refractory status epilepticus patients. Brain Dev. 2019 Sep;41(8):740. doi: 10.1016/j.braindev.2019.02.008. Epub 2019 Feb 22. No abstract available. PMID 30803732
- [Background] Cervenka MC, Henry BJ, Felton EA, Patton K, Kossoff EH. Establishing an Adult Epilepsy Diet Center: Experience, efficacy and challenges. Epilepsy Behav. 2016 May;58:61-8. doi: 10.1016/j.yebeh.2016.02.038. Epub 2016 Apr 6. PMID 27060389
- [Background] van der Louw EJ, Williams TJ, Henry-Barron BJ, Olieman JF, Duvekot JJ, Vermeulen MJ, Bannink N, Williams M, Neuteboom RF, Kossoff EH, Catsman-Berrevoets CE, Cervenka MC. Ketogenic diet therapy for epilepsy during pregnancy: A case series. Seizure. 2017 Feb;45:198-201. doi: 10.1016/j.seizure.2016.12.019. Epub 2016 Dec 26. PMID 28110175
- [Background] Kossoff EH, Zupec-Kania BA, Auvin S, Ballaban-Gil KR, Christina Bergqvist AG, Blackford R, Buchhalter JR, Caraballo RH, Cross JH, Dahlin MG, Donner EJ, Guzel O, Jehle RS, Klepper J, Kang HC, Lambrechts DA, Liu YMC, Nathan JK, Nordli DR Jr, Pfeifer HH, Rho JM, Scheffer IE, Sharma S, Stafstrom CE, Thiele EA, Turner Z, Vaccarezza MM, van der Louw EJTM, Veggiotti P, Wheless JW, Wirrell EC; Charlie Foundation; Matthew's Friends; Practice Committee of the Child Neurology Society. Optimal clinical management of children receiving dietary therapies for epilepsy: Updated recommendations of the International Ketogenic Diet Study Group. Epilepsia Open. 2018 May 21;3(2):175-192. doi: 10.1002/epi4.12225. eCollection 2018 Jun. PMID 29881797
- [Background] Correction to Lancet Respir Med 2020; published online Feb 21. https://doi.org/10.1016/S2213-2600(20)30079-5. Lancet Respir Med. 2020 Apr;8(4):e26. doi: 10.1016/S2213-2600(20)30103-X. Epub 2020 Feb 28. No abstract available. PMID 32119827
- See also: Severe Outcomes Among Patients with Coronavirus Disease 2019 (COVID-19) - United States, February 12-March 16, 2020 — https://www.cdc.gov/mmwr/volumes/69/wr/mm6912e2.htm